CLINICAL TRIAL: NCT04013061
Title: Impact of a Pharmacist-anesthesiologist Collaboration During Anesthesia Consultation on Prevention of Perioperative Medication Errors of Patients in Programmed Surgery
Acronym: PREVEMCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PHRCI/2018/GL-01
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2022-03

CONDITIONS: Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard consultation (No Intervention)
- Pharmacist-anesthesiologist consultation (Experimental)
  Interventions: Other: Pluridisciplinary consultation

INTERVENTIONS:
Other: Pluridisciplinary consultation — Pharmacist-anesthesiologist team will be present during the anesthetic consultation
  Arms: Pharmacist-anesthesiologist consultation

SUMMARY:
The investigators will evaluate the efficiency of a pharmacist-anesthesiologist collaboration in the anesthetic consultation in the prevention of medical errors perioperatively in patients undergoing scheduled surgery

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent
* The patient must be a member or beneficiary of a health insurance plan
* The patient has at least one chronic medication prescription (associated with a chronic illness)
* The patient is hospitalized for a programmed surgery in the service of urology or digestive surgery at the CHU Nimes or orthopedic surgery in the CHU Montpellier or Toulouse

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is having ambulatory programmed surgery
* The patient has an anesthetic consultation in a different health establishment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of patients with at least one medication error for chronic treatment | 48 hours post-admission
  %

SECONDARY OUTCOMES:
Nature of medication error | 48 hours post-admission
  According to REMED (Revue des Erreurs liées aux Médicaments Et Dispositifs médicaux) classification
Rate of medication errors corrected | 48 hours post-admission
  %
Rate of prescriptions respecting the Société Française d'Anesthésie et de Réanimation recommendations | 48 hours post-admission
  %
Rate of corrected medication errors or major, critical or catastrophic severity according to HAS 2018 | 48 hours post-admission
  %
Rate of patients whose usually prescribed medication at admission is not available for them in the evening following surgery | 48 hours post-admission
  %
Rate of medications not available on the establishment's therapeutic book and not brought by the patient | 48 hours post-admission
  %
Duration in hospital | End of hospitalization (max 30 days)
  Days
Rate of delay or cancellation of surgery linked to preoperational medication error | End of study (13 months)
  %

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine Leguelinel-Blache, Study Director — CHU Nimes
Locations (3):
- France (3):
  - CHU de Montpellier, Montpellier
  - CHU de Nimes, Nîmes
  - CHU de Toulouse, Toulouse